CLINICAL TRIAL: NCT03477201
Title: Characterizing Stray Energy Injuries During Robotic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-0527
Record Dates: First submitted 2018-03-09; First posted 2018-03-26 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Port-site Injury Caused by Stray Energy Transfer

STUDY DESIGN:
Intervention Model Description: The investigators plan to conduct a prospective, randomized controlled trial of patients undergoing elective laparoscopic or robotic unilateral inguinal hernia repair. Patients will be randomized into two groups, with one group undergoing laparoscopic transabdominal preperitoneal (TAPP) technique and a second group undergoing robotic inguinal hernia repair (TAPP technique) with the Xi DaVinci System (Intuitive, Sunnyvale, CA). The monopolar instrument will deliver via standard instruments on 30W coagulation mode (ForceTriad electrosurgical generator, Covidien, Boulder, CO). At the completion of the procedure, skin biopsies will be taken at each of the three port incisions. These samples will be examined for visual and histologic evidence of thermal injury by a blinded pathologist.
Who Masked: Participant
Masking Description: Patients will be randomized into two groups either laparoscopic or robotic assisted arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic robotic DaVinci assisted inguinal hernia repair (Experimental): Intervention: 30 patients will undergo a robotic assisted laparoscopic inguinal hernia repair. This will be done using the DaVinci Robotic Platform by Intuitive Surgical. This an accepted safe method of repairing inguinal hernia. This platform uses special robotic ports produced and supplied by Intuitive Surgical required to dock the machine to the patient. Monopolar energy will be provided by a ForceTriad system (Covidien, Boulder, CO), standard an common system used in most ORs. This will be used for dissection. The investigators will obtain small biopsies from port site to assess stray energy transfer injury, a model described by earlier studies.
  Interventions: Procedure: Laparoscopic robotic DaVinci assisted inguinal hernia repair
- Standard Laparoscopic inguinal hernia repair (Active Comparator): Intervention: 30 patients will undergo a laparoscopic inguinal hernia repair, an accepted safe method of repairing inguinal hernia. This platform uses standard laparoscopic ports. In our institution we use plastic ports made by Covidien, Boulder, CO. The operation will require two 5mm VersaPort (Covidien) and a Hassan Port. As in the robotic arm, monopolar energy will be provided by a ForceTriad system (Covidien, Boulder, CO), standard an common system used in most ORs. This will be used for dissection. The investigators will obtain small biopsies from port site to assess stray energy transfer injury, a model described by earlier studies.
  Interventions: Procedure: Standard laparoscopic inguinal hernia repair

INTERVENTIONS:
Procedure: Laparoscopic robotic DaVinci assisted inguinal hernia repair — Laparoscopic inguinal hernia repair using a robotic assisted laparoscopic procedure.
  Other Names: Dissection use of monopolar energy provided bt ForceTriad System (Covidien)
  Arms: Laparoscopic robotic DaVinci assisted inguinal hernia repair
Procedure: Standard laparoscopic inguinal hernia repair — Laparoscopic inguinal hernia repair, an accepted safe method of repairing inguinal hernia.
  Other Names: Dissection use of monopolar energy provided by ForceTriad System (Covidien)
  Arms: Standard Laparoscopic inguinal hernia repair

SUMMARY:
Stray energy transfer during laparoscopic surgery is recognized as a cause of potentially serious complications. This will be the first study to demonstrate clinical evidence of tissue injury due to stray energy transfer during robotic surgery. This information can then be used to define surgeon modifiable factors that can reduce the risk of patient injury. In addition, these data can guide the development of future robotic and laparoscopic platforms.

DETAILED DESCRIPTION:
BACKGROUND: Stray energy transfer from monopolar instruments during laparoscopic surgery is recognized as a cause of potentially catastrophic complications. The investigators have published multiple studies on the varied mechanisms of stray energy transfer during laparoscopic procedures. In addition, a preliminary study by the investigators has confirmed stray energy transfer during robotic surgery in an in vivo model. However, there are no data available on the potential clinical impact of stray energy in robotic surgery. Furthermore, there are no studies directly comparing stray energy transfer between laparoscopic and robotic procedures.

PURPOSE: The purpose of this study is to assess for thermal injury due to stray energy transfer during elective laparoscopic and robotic inguinal hernia repairs.

HYPOTHESIS: The Investigators hypothesize that thermal injury to the skin surrounding the working ports occurs during robotic and laparoscopic procedures. Based on prior data, the Investigators hypothesize these injuries will occur more frequently at the camera port during laparoscopy, and at the assistant port during robotic surgery.

METHODS: The Investigators plan to conduct a prospective, randomized controlled trial of patients undergoing elective laparoscopic or robotic unilateral inguinal hernia repair. Patients will be randomized into two groups, with one group undergoing laparoscopic transabdominal preperitoneal (TAPP) technique and a second group undergoing robotic inguinal hernia repair (TAPP technique) with the Xi DaVinci System (Intuitive, Sunnyvale, CA). The monopolar instrument will deliver via standard instruments on 30W coagulation mode (ForceTriad electrosurgical generator, Covidien, Boulder, CO). At the completion of the procedure, skin biopsies will be taken at each of the three port incisions. These samples will be examined for visual and histologic evidence of thermal injury by a blinded pathologist.

IMPORTANCE: This will be the first study to demonstrate clinical evidence of tissue injury due to stray energy transfer during robotic surgery. The inclusion of a laparoscopic arm will allow confirmation of prior study findings as well as direct comparison of stray energy transfer in both modalities. This information can then be used to define surgeon modifiable factors that can reduce the risk of patient injury. In addition, these data can guide the development of future robotic and laparoscopic platforms.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited in the general surgery clinic once the presence of an operable, inguinal hernia has been identified.
* All patients with a unilateral, symptomatic, inguinal hernia, and
* Who are surgical candidates for a laparoscopic inguinal hernia repair.

Exclusion Criteria:

* Under 18 years,
* Emergent hernia repairs,
* Recurrent hernias,
* Bilateral hernias, and
* Incarcerated bowel.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Most of inguinal hernia patients, especially at the VA are male and inguinal hernia is a different operation in female patients, thus male patients only will be included.
Enrollment: 42 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Histologic analysis of port-site skin biopsies | Biopsies will be taken right away and analysed within 1-2 weeks.
  Samples will be taken at the time of surgery from each of the three ports and analyzed by a board certified pathologist to assess for injury on histologic level.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Wikiel, MD, Principal Investigator — ECHCS/Denver VA
Locations (1):
- RMR Denver VA, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.